CLINICAL TRIAL: NCT03726749
Title: Tocilizumab Plus a Short Prednisone Taper for Giant Cell Arteritis (GCA)
Brief Title: Tocilizumab Plus a Short Prednisone Taper for GCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Principal Investigator, Sebastian H Unizony, MD, Assistant Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML40859
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Giant Cell Arteritis
Keywords: GCA; Tocilizumab; Prednisone
MeSH Terms: conditions — Giant Cell Arteritis | interventions — tocilizumab; Prednisone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tocilizumab and prednisone (Experimental): 1. TCZ 162 mg administered by subcutaneous injection weekly for 52 weeks.
  2. Prednisone taper over 8 weeks with a starting dose between 20 and 60 mg.
  Interventions: Drug: Tocilizumab; Drug: Prednisone

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab is an interleukin-6 (IL-6) receptor inhibitor
  Other Names: ACTEMRA®
Drug: Prednisone — Prednisone is an anti-inflammatory medication
  Other Names: Glucocorticoids

SUMMARY:
This is an open-label pilot study of tocilizumab (TCZ) 162 mg weekly administered subcutaneously for 52 weeks in combination with 8 weeks of oral prednisone.

DETAILED DESCRIPTION:
This is a single center, open label study that will assess the efficacy and safety of 52 weeks of tocilizumab (TCZ) in combination with 8-weeks of prednisone in 30 patients with active giant cell arteritis (GCA). Active disease is defined as signs and/or symptoms of GCA plus increased inflammatory markers (e.g., erythrosedimentation rate [ESR] and/or C-reactive protein [CRP]).

The study will enroll subjects with new onset and with relapsing/refractory GCA, and consist of a screening phase (up to 6 weeks), a treatment phase (52 weeks) and a safety follow up phase (4 weeks).

The primary endpoint of the study, sustained remission, will be assessed at week 52.

The definition of sustained remission contains 3 elements:

1. Absence of clinical signs and symptoms of active GCA along with the normalization of the ESR (< 40 mm/hour) and CRP (< 10 mg/L).
2. Completion of the pre-specified prednisone taper protocol
3. Absence of disease flare (relapse) since the induction of remission by week 8.

Disease flare is defined as the re-appearance of unequivocal signs or symptoms of active GCA (with or without elevation of ESR and/or CRP) or the elevation of the ESR and/or CRP that is thought to be due to active GCA and that requires escape therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent and to comply with the study protocol
2. Diagnosis of GCA classified per the following criteria:

   • Age 50 years or older

   AND at least one of the following:
   * Unequivocal cranial symptoms of GCA (new-onset localized headache, scalp tenderness, temporal artery tenderness or decreased pulsation, ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication)
   * Symptoms of polymyalgia rheumatica (PMR), defined as shoulder and / or hip girdle pain associated with inflammatory morning stiffness

   AND at least one of the following:
   * Cranial artery biopsy revealing features of GCA (e.g., mononuclear cell infiltration or granulomatous inflammation).
   * Evidence of large-vessel vasculitis by angiography or cross-sectional imaging study such as Image result for magnetic resonance angiogram (MRA), Computed tomography angiography (CTA) , or Image result for positron emission tomography (PET) and computed tomography (CT) (PET-CT)
   * Ultrasound demonstration of features of GCA in a cranial artery.
3. New-onset or relapsing/refractory active disease defined as follows:

   * New onset: diagnosis of GCA within 6 weeks of baseline visit
   * Relapsing/refractory: diagnosis of GCA > 6 weeks before baseline visit

AND

• Active GCA within 6 weeks of baseline visit defined as the presence of clinical signs and symptoms [cranial or PMR] and erythrocyte sedimentation rate (ESR) ≥ 30 mm/hour or C-reactive protein (CRP) ≥ 10 mg/L)

Exclusion Criteria:

1. General exclusion criteria

   * Major surgery within 8 weeks prior to screening or planned major surgery within 12 months after randomization
   * Transplanted organs (except corneal transplant performed more than 3 months prior to screening)
   * Major ischemic event, unrelated to GCA, within 12 weeks of screening
2. Exclusions related to prior or concomitant therapy*

   * Treatment with any investigational agent within 12 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
   * Previous treatment with cell-depleting therapies, including investigational agents, including but not limited to Campath (alemtuzumab), anti-CD4 (cluster of differentiation 4), anti-CD5, anti-CD3, anti-CD19, and anti-CD20
   * Previous treatment with alkylating agents, such as chlorambucil, or with total lymphoid irradiation
   * Immunization with a live/attenuated vaccine within ≤ 4 weeks prior to baseline
   * Treatment with cyclosporine A, azathioprine, cyclophosphamide or Mycophenolate mofetil (MMF) within 4 weeks of baseline. Patients on methotrexate at screening will require discontinuation of this agent prior to baseline visit.
   * Treatment with etanercept within 2 weeks; infliximab, certolizumab, golimumab, abatacept, or adalimumab within 8 weeks; or anakinra within 1 week of baseline
   * Patients requiring systemic glucocorticoid therapy for conditions other than GCA, which, in the opinion of the investigator, would interfere with adherence to the fixed glucocorticoid taper regimen and/or to assessment of efficacy in response to TCZ
   * Inability, in the opinion of the investigator, to withdraw GC treatment through protocol-defined taper regimen due to suspected or established adrenal insufficiency

     * Patients treated with TCZ before will be permitted to participate in the trial if they demonstrated treatment efficacy and they did not discontinue TCZ because of an adverse effect.
3. Exclusions related to general safety

   * History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies or to prednisone
   * Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus), psychiatric, osteoporosis/osteomalacia, glaucoma, corneal ulcers/injuries, or gastrointestinal (GI) disease
   * Current liver disease, as determined by the investigator
   * History of diverticulitis or active chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis, or other symptomatic lower GI conditions that might predispose a patient to perforations
   * Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis [TB] and atypical mycobacterial disease, hepatitis B and C, and herpes zoster, but excluding fungal infections of the nail beds)
   * Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
   * Active TB requiring treatment within the previous 3 years. Patients treated for TB with no recurrence within 3 years are eligible
   * Untreated latent TB infection (LTBI). Patients should be screened for latent TB and, if positive, treated according to local practice guidelines prior to initiating TCZ treatment. Patients treated for LTBI within 3 years are eligible. Patients with current LTBI are eligible for enrollment one month after initiating treatment for LTBI.
   * Primary or secondary immunodeficiency (history of or currently active)
   * Evidence of malignant disease or malignancies diagnosed within the previous 5 years (except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that have been excised and cured)
   * Females of childbearing potential and females who are breastfeeding
   * Males of reproductive potential who are not willing to use an effective method of contraception, such as condom, sterilization, or true abstinence throughout study and for a minimum of 6 months after study drug therapy
   * History of alcohol, drug, or chemical abuse within 1 year prior to screening
4. Laboratory exclusions

   * ALT or AST > 1.5 × upper limit of normal (ULN)
   * Total bilirubin > ULN
   * Platelet count < 100× 109/L (100,000/mm3)
   * Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
   * White blood cells < 3.0 × 109/L (3000/mm3)
   * Absolute neutrophil count < 1.0 × 109/L (1000/mm3)
   * Absolute lymphocyte count < 0.5 × 109/L (500/mm3)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana D Fernandes, MA, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unizony S, Matza MA, Jarvie A, O'Dea D, Fernandes AD, Stone JH. Treatment for giant cell arteritis with 8 weeks of prednisone in combination with tocilizumab: a single-arm, open-label, proof-of-concept study. Lancet Rheumatol. 2023 Dec;5(12):e736-e742. doi: 10.1016/S2665-9913(23)00265-5. Epub 2023 Nov 2. PMID 38251564

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab and Prednisone: 1. TCZ 162 mg administered by subcutaneous injection weekly for 52 weeks.
  2. Prednisone taper over 8 weeks with a starting dose between 20 and 60 mg.
  Tocilizumab: Tocilizumab is an interleukin-6 (IL-6) receptor inhibitor
  Prednisone: Prednisone is an anti-inflammatory medication
Period: Overall Study
Arm/Group | Tocilizumab and Prednisone
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab and Prednisone
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Sustained Remission
Description: Number and percentage of patients in sustained remission by week 52. Sustained remission was defined as the absence of disease flare between baseline and week 52. Flare was defined as the re-appearance of clinical manifestations of GCA with or without elevation of the inflammatory makers erythrocyte sedimentation rate (ESR) and/or C-reactive protein (CRP)
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab and Prednisone
Number analyzed (Participants) | 30
Participants | 23

2. Secondary Outcome: Disease Flares
Description: Total number of disease flares by week 52. Flare was defined as the re-appearance of clinical manifestations of GCA with or without elevation of the inflammatory makers erythrocyte sedimentation rate (ESR) and/or C-reactive protein (CRP)
Time Frame: 52 Weeks
Measure: Number; unit: Total number of flares
Arm/Group | Tocilizumab and Prednisone
Number analyzed (Participants) | 30
Total number of flares | 9

3. Secondary Outcome: Cumulative Prednisone Dose
Description: Cumulative prednisone dose (mg) by week 52
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tocilizumab and Prednisone
Number analyzed (Participants) | 30
mg | 1187 (470.4)

4. Secondary Outcome: Adverse Events
Description: Number and percentage of participants with at least one adverse event by week 52
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Tocilizumab Plus Prednisone Treatment: TCZ 162 mg administered by subcutaneous injection weekly for 52 weeks.
  Prednisone taper over 8 weeks with a starting dose between 20 and 60 mg.
Arm/Group | Tocilizumab Plus Prednisone Treatment
Number analyzed (Participants) | 30
Participants | 30

5. Secondary Outcome: Serious Adverse Events
Description: Number and percentage of participants with at least one serious adverse event by week 52
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab and Prednisone
Number analyzed (Participants) | 30
Participants | 4

ADVERSE EVENTS:
Time Frame: 2.2 years
Arm/Group | Tocilizumab and Prednisone
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab and Prednisone (N=30)
Olecranon bursitis, septic (Infections and infestations) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Osteoporotic vertebral fracture (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT03726749/Prot_SAP_002.pdf